CLINICAL TRIAL: NCT06524986
Title: The Effect of Self-Efficacy Promoting Program Using Computer Game on Proteinuria in Thai Children With Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Suwimon Rojnawee, PhD, RN, Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0814/65
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Nephrotic Syndrome; Proteinuria; School-Age Children; Self-Efficacy; Computer Game
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria

STUDY DESIGN:
Intervention Model Description: The experimental group underwent a program that aimed to enhance self-efficacy through computer games for a duration of 5 weeks, whereas the control group received regular nursing care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-efficacy promoting program (Experimental): The self-efficacy promotion program, inspired by Bandura's principles (1997, 2001) and employing computer games, extends across 5 weeks with 30-minute sessions conducted 10 minutes.The program involved activities such as motivation, modeling, and enactive mastery experiences. Weekly sessions covered collaborative planning, video demonstrations, interactive gaming, and follow-up calls to ensure active participation and address concerns related to physiological and affective states.
  Interventions: Behavioral: Self-efficacy promoting program using computer game
- Standard nursing care (Experimental): The control group received standard nursing care, which included providing dietary recommendations for pediatric patients. The recommended daily intake consisted of 0.8 grams of protein per kilogram of the child's weight, low-sodium foods, and low-fat options. This personalized guidance was communicated through informational brochures.
  Interventions: Behavioral: Standard nursing care

INTERVENTIONS:
Behavioral: Self-efficacy promoting program using computer game — The self-efficacy promotion program, inspired by Bandura's principles (1997, 2001) and employing computer games, extends across 5 weeks with 30-minute sessions conducted 10 minutes. Activities include: 1) Enactive Mastery Experiences 2) Modeling 3) Verbal Persuasion 4) Physiological and Affective States Assessment
  Arms: Self-efficacy promoting program
Behavioral: Standard nursing care — The control group received standard nursing care, which included providing dietary recommendations for pediatric patients. The recommended daily intake consisted of 0.8 grams of protein per kilogram of the child's weight, low-sodium foods, and low-fat options. This personalized guidance was communicated through informational brochures.
  Arms: Standard nursing care

SUMMARY:
Nephrotic syndrome is a medical condition where the kidneys release substantial amounts of protein into the urine, resulting in various issues such as tissue swelling and an increased susceptibility to infections. Emphasizing the importance of adequate nutrition and symptom monitoring is crucial in managing urine protein levels and mitigating associated complications.

The purpose of this study was to boost self-efficacy through a computer game-based program, aiding pediatric patients with Nephrotic syndrome in the adoption of healthy eating habits and efficient management of urine protein levels.

DETAILED DESCRIPTION:
This study was Quasi-experimental Research. Two group pre-test post-test with repeated measures design. Forty school-age children diagnosed with nephrotic syndrome were randomly allocated into two groups, with the participants distributed between an experimental group and a control group, each comprising 20 individuals. The experimental group underwent a program that aimed to enhance self-efficacy through computer games for a duration of 5 weeks, whereas the control group received regular nursing care. Information was gathered through personal record forms, urine protein assessments with test strips, dietary behavior surveys for school-age children with nephrotic symptoms, and self-efficacy surveys related to dietary behavior within the same group. The data underwent analysis using repeated measures analysis of variance. Statistical significance was defined as p < .05.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of nephrotic syndrome diagnosis by a physician and continuous hospital treatment for a minimum of 3 months.
* Presence of proteinuria levels at 1+ or higher during morning awakening or a urine protein quantity exceeding 30 mg/dL within the past 6 months (verified through medical records).
* Proficient communication skills in the Thai language.
* Ownership of a telephone or device suitable for gaming and internet connectivity.
* Willingness and cooperation from both the family and the child to actively participate in the research.
* Discontinuation of steroid medication by school-age patients.

Exclusion Criteria:

* involve symptoms indicative of a critical condition, such as entering a crisis or severe complications like heart failure or pleural effusion.
* school-age patients whose treatment plan has been modified by a physician, including the use of injectable medication instead of oral drugs or those receiving treatment in an inpatient setting.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Protein levels in the urine | Change from Baseline Protein levels in the urine at 5 weeks, followed by three days of consecutive follow-up calls
  Urine dipstick test assessments with COMBI-SCREEN® GP test strips

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Rojnawee, Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Nursing, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leddy J, Green JA, Yule C, Molecavage J, Coresh J, Chang AR. Improving proteinuria screening with mailed smartphone urinalysis testing in previously unscreened patients with hypertension: a randomized controlled trial. BMC Nephrol. 2019 Apr 18;20(1):132. doi: 10.1186/s12882-019-1324-z. PMID 30999886
- [Result] Jari M, Merrikhi A, Kelishadi R, Ghaffarzadeh Z. The First Report on the Frequency of Asymptomatic Proteinuria in Iranian School-aged Children. Adv Biomed Res. 2018 Feb 21;7:35. doi: 10.4103/2277-9175.225923. eCollection 2018. PMID 29531933
- [Result] Kato-Lin YC, Kumar UB, Sri Prakash B, Prakash B, Varadan V, Agnihotri S, Subramanyam N, Krishnatray P, Padman R. Impact of Pediatric Mobile Game Play on Healthy Eating Behavior: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 18;8(11):e15717. doi: 10.2196/15717. PMID 33206054
- [Result] Mishra R, Kumari S, Pathak A, Prasad KN, Malakar J. Risk factors for relapse in pediatric nephrotic syndrome in Ranchi. J Family Med Prim Care. 2023 Feb;12(2):223-226. doi: 10.4103/jfmpc.jfmpc_983_22. Epub 2023 Feb 28. PMID 37090998
- [Result] Downie ML, Gallibois C, Parekh RS, Noone DG. Nephrotic syndrome in infants and children: pathophysiology and management. Paediatr Int Child Health. 2017 Nov;37(4):248-258. doi: 10.1080/20469047.2017.1374003. Epub 2017 Sep 15. PMID 28914167
- [Result] Esezobor C, Ademola AD, Adetunji AE, Anigilaje EA, Batte A, Jiya-Bello FN, Furia FF, Muoneke U, McCulloch M, Nourse P, Obiagwu P, Odetunde O, Okyere P, Solarin A, Tannor EK, Noone D, Gbadegesin R, Parekh RS; Human Hereditary and Health in Africa Kidney Disease Research Network. Management of idiopathic childhood nephrotic syndrome in sub-Saharan Africa: Ibadan consensus statement. Kidney Int. 2021 Jan;99(1):59-67. doi: 10.1016/j.kint.2020.07.045. Epub 2020 Aug 29. No abstract available. PMID 32866504